CLINICAL TRIAL: NCT04879719
Title: The Influence of Ego-depletion on Implicit Aggression and Cognitive Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Ego-depletion study
Record Dates: First submitted 2021-05-03; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Aggression
Keywords: ego-depletion; implicit aggression; word-stem completion task; implicit association task
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either a ego-depletion- or a control group.
Who Masked: Participant
Masking Description: Participants do not know that there exists more than one condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ego-depletion group (Experimental): Participants in this condition are asked to suppress their emotion while watching an emotional video of a surgery. Suppressing the natural emotional reaction to such a video demands cognitive resources and thus can induce a state of ego-depletion.
  Interventions: Behavioral: Ego-depletion
- Control group (Active Comparator): Participants in the control group are asked to watch the same emotional video. However, they are required to simply watch the video without suppressing any emotions.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Ego-depletion — The surgery video lasts for 9 minutes and participants are asked to suppress their emotions. After the intervention several implicit aggression tests, as well as a task, measuring cognitive performance in general are assessed.
  Arms: Ego-depletion group
Behavioral: Control — The surgery video lasts for 9 minutes and participants in the control group are asked to watch the surgery video without the need to suppress their emotions. Several implicit aggression tests, as well as a task, measuring cognitive performance in general are assessed after the 9 minute video sequence.
  Arms: Control group

SUMMARY:
The aim of the planned online study is twofold. First, it opts to deliver further evidence for the existence of the construct ego-depletion. Second, it tries to further validate the German version of the word-stem completion task as a measure of implicit aggression. The psychological assessment of aggression is not a trivial aspect, however. In general, explicit measures of aggression have a higher face validity than their implicit counterparts. However, even implicit measures, such as the implicit association test for aggression, have a certain amount of face validity, since participants might be able to infer that the task is related to aggression. Another implicit aggression measure is the word-stem completion task, which asks participants to complement word-stems in order to build words. Lately, we have developed a German version of this task and found some promising first results, i.e., a factor analysis indicated that the word-stem completion task explained unique variance in aggression. The present study aims to further validate the German version of the word-stem completion task by experimentally manipulating aggression through an ego-depletion paradigm, in which cognitive resources are depleted. It is expected that participants in the ego-depletion condition build more aggressive solutions on the word-stem completion task than participants in the control group.

DETAILED DESCRIPTION:
Almost every one of us knows the experience of falling short of one's own resolutions, despite having the intention to behave differently. In dual-process models human behavior is proposed to be a result of reciprocal activity of an impulsive and a reflective system with the impulsive system being fast, associative, and mostly unconscious, while the activity of the reflective system is slow, rule-based and relies on cognitive resources. Hence, people are more prone to rely on the associative system if cognitive resources are diminished or temporarily unavailable. Such a state of low mental resources has been linked to various detrimental effects such as impulse buying, stereotyping, unhealthy food choices, aggression, as well as impaired cognitive performance in general and is referred to as ego-depletion. According to ego-depletion theory self-control functions like a muscle and activities that heavily rely on the exertion of self-control successively exhaust this limited resource. Lately, some critical concerns questioning the magnitude of ego-depletion effects or its existence altogether have been raised. Most recent meta-analytical findings resolved most of the uncertainty, however, and stressed the importance of the paradigm used to deplete cognitive resources with emotion suppression videos being best suited to induce a state of ego-depletion.

Therefore, an emotional video, showing sequences of a surgery will be used in the present research in order to manipulate the amount of cognitive resources available. While participants in the experimental group are asked to suppress any emotions while watching the video, the control group is requested to simply watch the video attentively.

The word-stem completion task is an implicit aggression measure that asks participants to complement word-stems with the assumption being that the more aggressive solutions a person generates the more aggressive that person is.

The experiment will use a sequential-task paradigm with half of the 60 participants being randomly assigned to the ego-depletion condition. After watching the emotional video, participants in both groups will be requested to complete the word-stem completion task, an aggression implicit association test, as well as a multi-source interference task. Furthermore, trait aggression and the amount of subjective emotion, experienced while watching the video, will be assessed as potential moderators.

It is expected that participants in the ego-depletion group will score higher on implicit aggression measures (word-stem completion task and implicit association task) and perform worse on the multi-source interference task, which measures cognitive performance.

Participants will be told that the experiment seeks to understand the relationship between emotional videos and cognition and creativity. At the end of the study, participants will be debriefed about the actual goal of the study and will receive monetary compensation for their participation.

ELIGIBILITY:
Inclusion Criteria:

* being mentally healthy
* German as native language
* being between 18-55 years in age

Exclusion Criteria:

* working in a medical profession

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-05-17 (Estimated); Study Completion 2021-05-17 (Estimated)

PRIMARY OUTCOMES:
Word-stem completion task | All measures will be taken on a single occasion in a sequential-task paradigm, which is standard in ego-depletion research. Completion of all tasks takes 6 minutes
  In the word-stem completion task participants are presented with up to 100 word-stems in random order. The participants' task is to build as many words as possible within sic minutes by complementing the word-stems. Solution words can be either aggressive, partially aggressive or non-aggressive. Sum scores for all aggressive and partially aggressive solutions are built as a first index of implicit aggression. First results from the German version of the word-stem completion task, however, indicate that a score taking into account the number of total solutions, as well as the word frequencies in the German language is better suited to measure implicit aggression than the conventional sum score method. Therefore, the new weighted score will be used as main outcome variable.
Implicit Association Test (IAT) for aggression | All measures will be taken on a single occasion in a sequential-task paradigm, which is standard in ego-depletion research. Completion of this task takes about 5 minutes.
  The IAT is a speeded classification task, which seeks to measure the inner strength of associations between certain concepts. During the IAT words are presented at the center of the screen and participants are asked to categorize stimuli either to the left or to the right based on the instructions of the respective block. IAT scores are obtained by comparing reaction times between blocks in which participants have to press the same button in response to aggressive as well as self-referential words with reaction times from blocks in which peaceful and self-referential words require the same response. If participants respond faster on trials in which aggressive and self-referential words require the same response this is thought to reflect higher levels of implicit aggression.
Multi-source interference task (MSIT) | All measures will be taken on a single occasion in a sequential-task paradigm, which is standard in ego-depletion research. Completion of this task takes about 5 minutes.
  The MSIT is thought to measure cognitive control and cognitive performance in general. On each trial three items are presented next to each other at the center of the screen, with two of them being identical and one deviating from the others. Participants are asked to identify the number that differs from the other two presented items (mostly numbers) and to press the corresponding key on the keyboard. The position and the actual number can either be the same, e.g. the number 2 presented in between two other numbers or letters (so-called flankers), in which we speak of congruency or number and position can be incongruent, for instance the number 2 presented left to

CONTACTS AND LOCATIONS:
Overall Officials: Simone Kühn, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Clinic Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumeister RF, Bratslavsky E, Muraven M, Tice DM. Ego depletion: is the active self a limited resource? J Pers Soc Psychol. 1998 May;74(5):1252-65. doi: 10.1037//0022-3514.74.5.1252. PMID 9599441
- [Background] Dang J. An updated meta-analysis of the ego depletion effect. Psychol Res. 2018 Jul;82(4):645-651. doi: 10.1007/s00426-017-0862-x. Epub 2017 Apr 8. PMID 28391367
- [Background] Hagger MS, Wood C, Stiff C, Chatzisarantis NL. Ego depletion and the strength model of self-control: a meta-analysis. Psychol Bull. 2010 Jul;136(4):495-525. doi: 10.1037/a0019486. PMID 20565167
- [Background] Strack F, Deutsch R. Reflective and impulsive determinants of social behavior. Pers Soc Psychol Rev. 2004;8(3):220-47. doi: 10.1207/s15327957pspr0803_1. PMID 15454347